CLINICAL TRIAL: NCT06904157
Title: Investigation of Shoulder Head Position, Upper Extremity Proprioception, and Upper Extremity Function in Adolescents With Idiopathic Scoliosis Using Braces
Brief Title: Investigation of Shoulder Position, Upper Extremity Proprioception, and Function in Adolescents With Idiopathic Scoliosis Using Braces
Status: Not yet recruiting | Type: Observational
Sponsor: Gözde Yagci (Gür) (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Gözde Yagci (Gür), Prof. Dr., Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: HU-KNurdogan-001; SBA 23/116 (Other: Hacettepe University Research Ethics Committee)
Record Dates: First submitted 2025-02-27; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Scoliosis; Brace; Upper Extremity; Proprioception; Function
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient Group: This group consists of individuals diagnosed with adolescent idiopathic scoliosis (AIS) who are using Cheneau-type braces. The age range for this group is 10-18 years. Participants must have a diagnosis of AIS, have been using a Cheneau-type brace for at least one month, have a primary thoracic or thoracolumbar curve, and a Cobb angle of 20 degrees or more. Additionally, the dominant hand must be the right hand, and participants must be willing to participate in the study with parental consent. Exclusion criteria include a diagnosis of congenital scoliosis, being a professional athlete, having a history of neuromuscular, rheumatological, renal, vestibular, pulmonary, or cardiovascular diseases unrelated to scoliosis, and a history of spinal surgery.
- Control Group: This group consists of healthy adolescents without any scoliosis or spinal deformities. The age range for this group is 10-18 years. Participants must have a dominant right hand and be willing to participate in the study. Exclusion criteria include a history of neuromuscular, rheumatological, renal, vestibular, pulmonary, or cardiovascular diseases, a history of spinal surgery, and being a professional athlete.

SUMMARY:
This study aims to investigate the effects of brace use on shoulder position, upper extremity proprioception, and upper extremity function in adolescents with idiopathic scoliosis. Participants will be assessed under both in-brace and out-brace conditions. The control group's upper extremity proprioception and upper extremity function will be assessed under out-brace condition. Shoulder position will be evaluated using a photographic method, while upper extremity proprioception (angular deviation) will be measured with the Laser Pointer-Assisted Angle Reproduction Test. Upper extremity function will be assessed through muscle strength tests, the Closed Kinetic Chain Upper Extremity Stability Test, the Medicine Ball Throw Test, the Finger-to-Nose Test, the Nellson Hand Reaction Test, and the Minnesota Manual Dexterity Test. Adolescents diagnosed with idiopathic scoliosis who have been prescribed brace treatment and have no history of spinal surgery or neurological/musculoskeletal conditions affecting upper extremity function will be included. Individuals with congenital or neuromuscular scoliosis, previous spinal surgery, neurological disorders affecting proprioception, or those unable to comply with study assessments will be excluded. This study aims to provide insights into the impact of bracing on proprioception and upper extremity function, contributing to the development of rehabilitation strategies for scoliosis management.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a complex three-dimensional spinal deformity characterized by lateral curvature and vertebral rotation, affecting postural alignment, musculoskeletal function, and neuromuscular control. AIS can lead to asymmetrical loading of the spine and trunk, potentially altering proprioception, postural stability, and functional capacity. Bracing is a widely used conservative treatment aimed at preventing curve progression and maintaining spinal alignment during skeletal growth. However, its effects on upper extremity function, proprioception, and shoulder biomechanics remain underexplored.

Proprioception, the body's ability to sense movement and position, plays a critical role in motor control and stability. In AIS, spinal asymmetry and altered postural alignment may disrupt proprioceptive feedback mechanisms, leading to compensatory movement strategies and potential impairments in upper extremity coordination and function. Additionally, bracing may impose external constraints that influence neuromuscular activation patterns and joint positioning, further affecting movement efficiency and functional performance.

This study aims to investigate the impact of brace use on shoulder position, upper extremity proprioception, and functional performance in adolescents with idiopathic scoliosis. Participants will be assessed in both braced and unbraced conditions to determine how brace-related mechanical constraints influence proprioceptive accuracy, postural adaptation, and functional motor skills. Shoulder position will be analyzed through photographic assessment, while proprioception will be measured using the Laser Pointer-Assisted Angle Reproduction Test. Upper extremity function will be evaluated using standardized clinical assessments, including strength tests, stability and coordination measures, and reaction time assessments.

Understanding the effects of bracing on upper extremity proprioception and function is essential for optimizing rehabilitation strategies in AIS. This study seeks to provide evidence that can inform clinical decision-making regarding brace design, therapy interventions, and functional training approaches to minimize movement restrictions and enhance musculoskeletal performance in adolescents undergoing brace treatment.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria for the patient group;

* To have a diagnosis of adolescent idiopathic scoliosis (AIS),
* Be using Cheneau Type corset for at least one month,
* Having a primary thoracic or thoracolumbar curve,
* Cobb angle of 20 degrees or more,
* The dominant hand is the right hand,
* Volunteering to participate in the study,
* Parental consent was required. Inclusion criteria for the control group;
* Individuals between the ages of 10-18
* Dominant Hand is the Right Hand
* Volunteering to Participate in the Study

Exclusion Criteria:

Exclusion Criteria for Patient Group;

* Having a diagnosis of Congenital Scoliosis,
* Becoming a Professional Athlete,
* Neuromuscular, Rheumatologic, Renal Except Scoliosis, Any History of Vestibular, Pulmonary or Cardiovascular Disease Finding
* History of Surgical Intervention on the Spine. Exclusion Criteria for Control Group;
* Neuromuscular, Rheumatologic, Renal, Vestibular, Pulmonary Or History of any Cardiovascular Disease
* History of Spine Surgery,
* Being a Professional Athlete.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will be carried out on adolescent idiopathic scoliosis individuals between the ages of 10-18 who have been using the brace prescribed by a physician for at least one month and age-matched healthy individuals. The corsets used by the individuals with scoliosis included in the study will be the previously prepared Cheneau type brace. Healthy individuals will be included in the study with the snowball method from the close environment of the individuals with scoliosis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle Measurement | Baseline and first week of brace use
  Cobb angle, a standard measurement used to quantify spinal curvature in scoliosis, will be obtained from physician notes and radiographic images. A tangent will be drawn along the superior edge of the uppermost involved vertebra and the inferior edge of the lowest involved vertebra. Perpendicular lines will then be drawn, and the angle at their intersection will be recorded. Cobb angle will be measured both with and without bracing, and the difference will be noted.
  Unit of Measure: Degrees (°)
Angle of Trunk Rotation (ATR) | Before brace application and 1 hour after brace application
  Trunk rotation will be assessed using a scoliometer during the Adams forward bending test. Participants will bend forward with arms hanging freely while the scoliometer will be placed perpendicularly on the spine and moved downward from the thoracic region. The highest degree of trunk rotation will be recorded.
  Unit of Measure: Degrees (°)
Upper Extremity Proprioception Accuracy | Before brace application and 1 hour after brace application
  Proprioception will be assessed using the Laser Pointer-Assisted Angle Reproduction Test (LPAART) at 55°, 90°, and 125° in shoulder flexion and abduction. A laser pointer will be attached to the dominant wrist, and participants will position their arm to the designated angle with eyes open. After memorizing the position, they will attempt to replicate it with eyes closed. The deviation from the target angle will be recorded.
  Unit of Measure: Degrees (°) of deviation
Anterior Humeral Head Position | Before brace application and 1 hour after brace application
  The anterior displacement of the humeral head relative to the acromion will be measured in two positions: (1) neutral shoulder position and (2) hands on hips (wrists extended, thumbs posterior). The distance between the anterior humeral head and the anterior acromion will be palpated, marked, photographed from 20 cm above, and measured in centimeters.
  Unit of Measure: Centimeters (cm)

SECONDARY OUTCOMES:
Upper Extremity Muscle Strength | Before brace application and 1 hour after brace application
  Isometric muscle strength of shoulder and elbow muscles will be assessed using a digital dynamometer (Power Track). Each test will be performed three times, and the highest value will be recorded in Newtons (N). Strength tests will include shoulder elevation (upper trapezius), flexion, abduction, internal and external rotation, elbow flexion, and extension.
  Unit of Measure: Newtons (N)
Hand Dexterity (Minnesota Dexterity Test) | Before brace application and 1 hour after brace application
  Hand dexterity will be assessed using the Minnesota Hand Dexterity Test, which includes two timed tasks: (1) placing disks in holes and (2) rotating disks. The total completion time will be recorded.
  Unit of Measure: Seconds (s)
Hand Reaction Time (Nelson Hand Reaction Test) | Before brace application and 1 hour after brace application
  Reaction time will be measured using the Nelson Hand Reaction Test, where participants will catch a dropped ruler between their thumb and index finger. The distance (cm) the ruler falls before being caught will be converted into reaction time using the formula: Reaction Time = √(2 × Distance / 980 ms²). The best and worst trials will be excluded, and the average of three trials will be recorded.
  Unit of Measure: Milliseconds (cm/ms)
Upper Extremity Coordination (Finger-to-Nose Test) | Before brace application and 1 hour after brace application
  Coordination will be assessed using the finger-to-nose test. Participants will touch their nose and then the examiner's finger, repeating the movement for 20 seconds. The number of successful repetitions will be recorded.
  Unit of Measure: Repetitions in 20 seconds
Closed Kinetic Chain Upper Extremity Stability (CKCUES) Test | Before brace application and 1 hour after brace application
  Participants will perform alternating hand touches between two lines (30 cm apart) while in a modified push-up position. The total number of touches in 15 seconds will be recorded.
  Unit of Measure: Number of touches
Open Kinetic Chain Upper Extremity Power (Medicine Ball Throw Test) | Before brace application and 1 hour after brace application
  Upper extremity explosive power will be assessed using the Medicine Ball Throw Test. Participants, kneeling on a mat, will throw a 3-kg medicine ball forward using a chest pass motion. The distance from the starting point to the first contact point will be measured. The best of three trials will be recorded.
  Unit of Measure: Centimeters (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University / Orthotics and Biomechanics Unit, Ankara, altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided